CLINICAL TRIAL: NCT06024486
Title: Correlation of Fibrinogen to Albumin Ratio and C-reactive Protein to Albumin Ratio With Disease Activity in Juvenile Idiopathic Arthritis
Brief Title: Fibrinogen to Albumin Ratio and C-reactive Protein to Albumin Ratio in Juvenile Idiopathic Arthritis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maha Sayed Ibrahim Abdelrahman, principal investigator, Assiut University
Other Study IDs: Juvenile arthritis assiut u
Record Dates: First submitted 2023-08-14; First posted 2023-09-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- JIA cases: juvenile idiopathic arthritis cases
  Interventions: Diagnostic Test: fibrinogen to albumin ratio (AFR) and C-reactive protein to albumin ratio (CAR)
- CONTROL: age and sex matched healthy controls
  Interventions: Diagnostic Test: fibrinogen to albumin ratio (AFR) and C-reactive protein to albumin ratio (CAR)

INTERVENTIONS:
Diagnostic Test: fibrinogen to albumin ratio (AFR) and C-reactive protein to albumin ratio (CAR) — measurement of serum albumin, fibrinogen and CRP

SUMMARY:
The fibrinogen to albumin ratio (FAR) and C-reactive protein to albumin ratio (CAR) have emerged as useful biomarkers to predict systemic inflammation. The aim here is to investigate the relation between FAR/CAR and Juvenile arthritis disease activity score (JASDAS27) in Juvenile idiopathic arthritis (JIA)

DETAILED DESCRIPTION:
The JADAS27 includes a selected count of the following joints: cervical spine, elbows, wrists, metacarpophalangeal joints (from first to third), proximal interphalangeal joints, hips, knees and ankles.

ELIGIBILITY:
Inclusion Criteria:

* All juvenile idiopathic arthritis fulfilling the criteria of International League of Associations for Rheumatology (ILAR) and age and sex matched healthy subjects

Exclusion Criteria:

* Other systemic inflammatory or autoimmune disorders.
* History of corticosteroid medication in the last 6 months.
* Liver diseases.
* Malignancy.

Max Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All juvenile idiopathic arthritis fulfilling the criteria of International League of Associations for Rheumatology (ILAR) and age and sex matched healthy subjects.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
The fibrinogen to albumin ratio | 3 months
  measurement of serum fibrinogen and albumin
The CRP to albumin ratio | 3 MONTHS
  measurement of serum CRP and albumin
Correlation of fibrinogen to albumin and CRP to albumin ratios on one side with disease activity on the other side | 3 MONTHS
  correlation of these ratios with JADAS27